CLINICAL TRIAL: NCT05136170
Title: 4-week,Phase III, Multicenter, Double-masked Clinical Study to Evaluate Safety-efficacy of Cenegermin (Oxervate®) 20 mcg/mL Ophthalmic Solution vs Vehicle in Patients With Severe Sjogren's Dry Eye Treated With Cyclosporine A (PROTEGO-2).
Brief Title: Study to Evaluate Safety and Efficacy of Cenegermin (Oxervate®) vs Vehicle in Severe Sjogren's Dry Eye Disease
Acronym: PROTEGO-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NGF0221; 2021-003749-39 (EudraCT Number)
Record Dates: First submitted 2021-11-15; First posted 2021-11-29 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Dry Eye Disease
Keywords: Sjogren's dry eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — cenegermin

STUDY DESIGN:
Intervention Model Description: multicenter, double-masked, vehicle-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This was a double-blind study.The vials containing cenegermin (20 mcg/mL) or vehicle were identical in appearance, and the contents of the vials were indistinguishable. All staff directly involved in the analysis of study results remained masked to treatment assignments while the study was in progress. The blind was not broken for any patient during the study before the database lock.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cenegermin (Experimental): One drop of cenegermin 20 mcg/mL (rhNGF 20 mcg/mL), in the pharmaceutical form of ophthalmic sterile solution, was instilled in both eyes three times daily (TID), every six hours.
  Interventions: Drug: Cenegermin
- Vehicle (Placebo Comparator): In this arm one drop of vehicle was instilled in both eyes TID for 28 consecutive days.
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: Cenegermin — Oxervate®, an ophthalmic solution containing cenegermin 20 mcg/mL, which is a recombinant human Nerve Growth Factor (rhNGF); one drop of the test product will be instilled in both eyes three times daily (TID) for 28 consecutive days.
  Other Names: Oxervate®
  Arms: Cenegermin
Other: Vehicle — Vehicle was instilled with the same scheme of the test product
  Other Names: Placebo
  Arms: Vehicle

SUMMARY:
Primary Objectives:

* To compare the efficacy of cenegermin vs vehicle in Schirmer I test (without anaesthesia) > 10 mm/5 min at Week 4 by testing the superiority.
* To compare the efficacy of cenegermin vs vehicle in Symptom Assessment in Dry Eye questionnaire (SANDE) global score at Week 12 by testing the superiority.

Secondary Objectives:

* To compare the efficacy of cenegermin vs vehicle in Schirmer I test at Week 4, 8, 12 and 16 by testing the superiority.
* To compare the efficacy of cenegermin vs vehicle in Cornea and conjunctiva vital staining with fluorescein (National Eye Institute [NEI] scales) at Week 4, 8, 12 and 16 by testing the superiority.
* To compare the efficacy of cenegermin vs vehicle in Tear Film Break-Up Time (TFBUT) at Week 4, 8, 12 and 16 by testing the superiority.
* To compare the efficacy of cenegermin vs vehicle in SANDE scores at Week 8, 12 and 16 by testing the superiority.
* To compare the efficacy of cenegermin vs vehicle in worsening in symptom scores (SANDE) and/or NEI score at Week 4 by testing the superiority.
* To compare the efficacy of cenegermin vs vehicle in impact of dry eye on everyday life (IDEEL) questionnaire at Week 4, 8, 12 and 16 by testing the superiority.

DETAILED DESCRIPTION:
This was a 4 week phase III, multicenter, double-masked, vehicle-controlled study to evaluate safety and efficacy of cenegermin ophthalmic solution at 20 mcg/mL solution versus vehicle, in patients with severe Sjogren's dry eye disease under treatment with Ciclosporine A (or other drugs of the same class).

During the Screening all procedures for inclusion and exclusion were performed. From the day of screening, the patients stopped any kind of further treatment, except CsA and commercially available preservative-free artificial tears provided by the Sponsor for a period of 8 days and 10 days as maximum. At the end of the washout period, patients still meeting the entry criteria for this study were randomized 1:1 and treated for 4 weeks with either cenegermin ophthalmic solution 20 mcg/mL three times a day (TID) or vehicle TID.

In addition to topical CsA eye drops (both groups continued with topical CsA eye drops, or other topical ophthalmic treatment of the same class), during the 4 weeks of masked treatment, only the administration of investigational medicinal product (IMP) was allowed.

During the follow up period, the patient could administer additional preservative-free artificial tear eye drops, provided by the Sponsor, only if strictly needed, and had to document in the patient's Diary the number of additional drops administered for each eye.

Patients were then followed-up for efficacy and safety endpoints until Week 16 and for safety endpoints until Week 24.

The total duration of the study was 25 weeks including 1 week of screening.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 18 years.
2. Patients with a confirmed diagnosis of Sjögren's syndrome or other autoimmune disease known to induce Sjögren's DED.
3. Patients with severe Sjögren's DED characterized by the following clinical features:

   1. Corneal and/or conjunctival staining with fluorescein using National Eye Institute (NEI) grading system ≥ 3.
   2. SANDE questionnaire >25 mm.
   3. Schirmer test I (without anaesthesia) ≥ 2 ≤ 5 mm/5 min.
4. The same eye (eligible eye) must fulfil all the above criteria.
5. Patients diagnosed with severe Sjögren's DED at least 3 months before enrolment (current use or recommended use of artificial tears for the treatment of Sjögren's related DE).
6. Best corrected distance visual acuity (BCDVA) score of ≥ 0.1 decimal units (20/200 Snellen value) in each eye at the time of study enrolment.
7. If a female of childbearing potential, have a negative urine pregnancy test and use a highly effective method to avoid pregnancy for the duration of the trial and 30 days after the study treatment period. Males of reproductive potential should use effective contraception during treatment and 30 days after the study treatment period.
8. Patients who have given written informed consent before any study-related procedures not part of standard medical care are performed.
9. Patients must have the ability and willingness to comply with study procedures.
10. Patients under treatment with topical cyclosporine (CsA), or topical ophthalmic treatments of the same class for at least 30 days before Screening Visit (Day -8).

Exclusion Criteria:

1. Inability to speak and understand the local language sufficiently to understand the nature of the study, to provide written informed consent, and to allow the completion of all study assessments.
2. Evidence of an active ocular infection, in either eye.
3. Presence of any other ocular disorder or condition requiring topical medication during the entire duration of study in either eye.
4. History of severe systemic allergy or of ocular allergy (including seasonal conjunctivitis) or chronic conjunctivitis and/or keratitis other than dry eye.
5. Intraocular inflammation defined as Tyndall score > 0.
6. History of malignancy in the last 5 years.
7. Systemic disease not stabilized within 1 month before Screening Visit (e.g., diabetes with glycemia out of range, thyroid malfunction) or judged by the Investigator to be incompatible with the study (e.g., current systemic infections) or with a condition incompatible with the frequent assessment required by the study.
8. Patient had a serious adverse reaction or significant hypersensitivity to any drug or chemically related compounds or had a clinically significant allergy to drugs, foods, amide local anaesthetics or other materials including commercial artificial tears (in the opinion of the Investigator).
9. Females of childbearing potential (those who are not surgically sterilized or post-menopausal for at least 1 year) were excluded from participation in the study if they met any one of the following conditions:

   1. were currently pregnant or,
   2. had a positive result at the urine pregnancy test (Baseline/Day 1) or,
   3. intended to become pregnant during the study treatment period or,
   4. were breast-feeding or,
   5. were not willing to use highly effective birth control measures, such as: combined (oestrogen and progesterone containing) hormonal contraceptives associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, implantable, injectable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomised partner, sexual abstinence - during the entire course of and 30 days after the study treatment period.
10. Any concurrent medical condition, that in the judgment of the PI, might interfere with the conduct of the study, confound the interpretation of the study results, or endanger the patient's well-being.
11. Use of topical corticosteroids, lifitegrast, autologous serum tears in either eye during the study (previous use not an exclusion criteria but must be discontinued at the Screening Visit).
12. Contact lenses, True Tear device, moisture goggles, sutureless amniotic membrane or punctum plug use during the study (previous use not an exclusion criteria but must be discontinued at the Screening Visit).
13. History of drug addiction or alcohol abuse in the last 2 years.
14. Any prior ocular surgery (including refractive, palpebral and cataract surgery) if within 90 days before the Screening Visit.
15. Participation in a clinical trial with a new active substance during the past 3 months.
16. Participation in another clinical trial study at the same time as the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Mantelli, MD, Study Director — Dompé Farmaceutici
Locations (10):
- United States (7):
  - Lugene Eye Institute - Glendale Office, Glendale, California
  - The Johns Hopkins University, Baltimore, Maryland
  - Tufts University School of Medicine (TUSM) - New England Eye Center/Tufts Medical Center, Boston, Massachusetts
  - OCLI (Ophthalmic Consultants of Long Island), Garden City, New York
  - Scheie Eye Institute, Philadelphia, Pennsylvania
  - Houston Eye Associates HEA - Gramercy Location, Houston, Tennessee
  - Toyos Clinic - Nashville, Nashville, Tennessee
- Italy (3):
  - AOU Gaspare Rodolico - Ospedale San Marco, Catania
  - Università degli Studi di Milano - Ospedale San Giuseppe - UO Oculistica, Milan
  - AOU Policlinico Umberto I - Dipartimento Organi di Senso - Clinica Oculistica, Roma

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three sites in Italy out of the four opened, and 7 sites in US enrolled patients. A total of 97 adult patients (≥ 18 years) with a diagnosis of severe Sjögren's DED was assessed for eligibility.
  There were 12 screening failures. The remaining patients (n=85) were randomized 1:1 as follows: 44 to cenegermin and 41 to vehicle. One patient in the vehicle group did not receive study medication and was excluded from the SAF and FAS.
Pre-assignment Details: No units other than participants were assigned.
Groups:
- Cenegermin: Oxervate®, an ophthalmic solution containing cenegermin 20 mcg/mL, which is a recombinant human Nerve Growth Factor (rhNGF). In this arm one drop of cenegermin 20 mcg/mL was instilled in both eyes TID for 28 consecutive days.
  Cenegermin: One drop of the test product was instilled in both eyes TID
- Vehicle: In this arm one drop of vehicle was a instilled in both eyes TID for 28 consecutive days.
  Vehicle: One drop of the placebo was instilled in both eyes TID
Period: Overall Study
Arm/Group | Cenegermin | Vehicle
Started | 44 | 41
Randomized But Not Treated | 0 | 1
Safety Population (SAF) | 44 | 40
Full Analysis Set Population (FAS) | 44 | 40
Per Protocol Set (PP) | 38 | 33
Completed | 41 | 39
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Can no longer make office visits | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis set (FAS): The FAS population consisted of all randomized patients who received at least one dose of the tnvestigational product. FAS population was analysed according to intention-to-treat (ITT) principle, i.e., by treatment allocation regardless happening of intercurrent events (treatment policy strategy). The FAS population was used for the primary analysis of the study and to present results on efficacy data.
Groups:
- Cenegermin - FAS: One drop of cenegermin 20 mcg/mL (rhNGF 20 mcg/mL), in the pharmaceutical form of ophthalmic sterile solution, was instilled in both eyes three times daily (TID), every six hours.
  Cenegermin: Oxervate®, an ophthalmic solution containing cenegermin 20 mcg/mL, which is a recombinant human Nerve Growth Factor (rhNGF); one drop of the test product will be instilled in both eyes three times daily (TID).
- Vehicle - FAS: In this arm one drop of vehicle was instilled in both eyes TID for 28 consecutive days.
  Vehicle: Vehicle was instilled with the same scheme of the test product
- Total: Total of all reporting groups
Arm/Group | Cenegermin - FAS | Vehicle - FAS | Total
Number analyzed (Participants) | 44 | 40 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 27 | 62
  >=65 years | 9 | 13 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (13.93) | 58.1 (12.84) | 56.5 (13.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 35 | 73
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 41 | 38 | 79
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 37 | 30 | 67
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42
  Italy | 23 | 19 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Schirmer I Test (Without Anesthesia) >10mm/5min in the Eligible Eye at Week 4
Description: The Schirmer test was used in ophthalmic examination to measure tear production for the diagnosis of conditions such as keratoconjunctivitis sicca and dry eye.
  Without previously instilling anesthetic drops, the Schirmer strip was inserted into the lower conjunctival sac at the junction of the lateral and middle thirds, avoiding touching the cornea, and the length of wetting strips in millimeters was recorded after 5 minutes.
  After 5 minutes had elapsed, the Schirmer's test strip was removed and the length of the tear absorption on the strip was measured (millimeters/5 minutes).
  Cutoff values:
  <5 mm - pathologic dry eye 5-10 mm - marginal dry eye >10 and <30 mm - normal secretion The longer, the wetted length, the healthier the status of the eye. No units other than participants were assigned.
Time Frame: At Week 4 (Visit 3)
Population: Full Analysis set The FAS population consisted of all randomized patients who received at least one dose of the investigational product. The FAS population was used for the primary analysis of the study and to present results on efficacy data. While at baseline FAS patients were n=44 for IMP and 40 for Vehicle, at week 4 patients analyzed were n=43 in the IMP group and n=39 in the Vehicle arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Cenegermin - FAS | Vehicle - FAS
Number analyzed (Participants) | 43 | 39
Participants | 19 | 4
Statistical Analysis 1: Comparison: Cenegermin - FAS vs Vehicle - FAS; Analysis was based on logistic regression model with multiple imputation (MI) under a missing not at random (MNAR) mechanism using retrieve dropouts with proportion of patients reaching a value of Schirmer I test > 10 mm/5 min at Week 4 as dependent variable, treatment, gender, age class and baseline Schirmer I test value as qualitative independent variables. Site was considered as random effects that vary randomly among patients; Test type: Superiority — The following null hypothesis was defined on this endpoint: the proportion of patients reaching a value of Schirmer I test (without anaesthesia) >10mm/5min at week 4 in cenegermin (rhNGF) was lower or equal than control. The null hypothesis was rejected if the associated primary analysis p-value was lower than 0.025; p = 0.002, Regression, Logistic — P-value of treatment variable from logistic regression model on proportion of patients reaching a value of Schirmer I test (without anesthesia) >10mm/5min; Odds Ratio (OR) = 8.498, 95% CI 2-sided [2.165 to 33.356]

2. Primary Outcome: Change From Baseline in Symptom Questionnaire (SANDE) Global Score at Week 12
Description: SANDE was a short questionnaire to evaluate both dry eye intensity and frequency. It uses a 100 mm horizontal line (Visual Analogue Scale - VAS), for each of the 2 questions, to assess ocular discomfort and/or dryness.
  Frequency of symptoms ranged from "rarely" (best outcome) to "all of the time" (worst outcome), while the severity of symptoms ranged from "very mild" (best outcome) to "very severe" (worst outcome). Patients had to place a mark on the two given lines based on the extent of their symptoms.
  The locations of the marks was measured in mm from left to right and recorded as frequency and severity scores, respectively.
  The SANDE lines for intensity and for severity ranged from 0, being the minimal amount of dry eye symptoms (best outcome) to 100, being the maximal amount of dry eye symptoms (worst outcome).
  The total SANDE score was calculated by multiplying the frequency score by the severity score and obtaining the square root (0-100; the lower, the better).
Time Frame: At Week 12 (Visit 5 - Follow up)
Population: Full Analysis set (FAS): The FAS population consisted of all randomized patients who received at least 1 dose of the IMP. The FAS population was used for the primary analysis of the study and to present results on efficacy data. No units other than participants were assigned.
  While at baseline FAS patients were n=44 for IMP and 40 for Vehicle, at week 12 patients analyzed were n=40 in the IMP group and n=39 in the Vehicle arm.
  Please note that mean is an adjusted mean.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cenegermin - FAS | Vehicle - FAS
Number analyzed (Participants) | 40 | 39
score on a scale | -12.452 [-19.962 to -4.942] | -13.042 [-20.650 to -5.433]
Statistical Analysis 1: Comparison: Cenegermin - FAS vs Vehicle - FAS; Analysis was based on ANCOVA model with multiple imputation (MI) under a missing not at random (MNAR) mechanism using retrieve dropouts with change from baseline in the global SANDE score at Week 12 as dependent variable, treatment, gender, age class and baseline global SANDE score as qualitative independent variables. Site was considered as random effects that vary randomly among patients; Test type: Superiority — The following null hypothesis is defined on this endpoint: the change from baseline (reduction) in the global SANDE score at week 12 in cenegermin is lower or equal than control. The null hypothesis is rejected if the associated primary analysis p-value is lower than 0.025; p = 0.890, ANCOVA — P-value of adjusted means difference between treatments from the ANCOVA model on change from baseline in the global SANDE score; Adjusted means difference = 0.59, 95% CI 2-sided [-7.801 to 8.981]

3. Secondary Outcome: Key Secondary Outcome: Number of Patients With Schirmer I Test (Without Anesthesia) >10mm/5min at Week 8
Description: The Schirmer test was used in ophthalmic examination to measure tear production for the diagnosis of conditions such as keratoconjunctivitis sicca and dry eye.
  Without previously instilling anesthetic drops, the Schirmer strip was inserted into the lower conjunctival sac at the junction of the lateral and middle thirds, avoiding touching the cornea, and the length of wetting strips in millimeters was recorded after 5 minutes.
  After 5 minutes had elapsed, the Schirmer test strip was removed and the length of the tear absorption on the strip was measured (millimeters/5 minutes).
  Cutoff values:
  <5 mm - pathologic dry eye 5-10 mm - marginal dry eye >10 and <30 mm - normal secretion The longer, the wetted length, the healthier the status of the eye. No units other than participants were assigned.
Time Frame: At Week 8 (Visit 4)
Population: Full Analysis set (FAS): The FAS population consisted of all randomized patients who received at least one dose of the investigational product. The FAS population was used for the primary analysis of the study and to present results on efficacy data. While at baseline FAS patients were n=44 for IMP and 40 for Vehicle, at week 8 patients analyzed were n=40 in the IMP group and n=38 in the Vehicle arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Cenegermin - FAS | Vehicle - FAS
Number analyzed (Participants) | 40 | 38
Participants | 11 | 2
Statistical Analysis 1: Comparison: Cenegermin - FAS vs Vehicle - FAS; This key secondary endpoint was analyzed by means of a logistic regression model with proportion of patients reaching a value of Schirmer I test >10mm/5min at Week 8 as dependent variable, treatment, gender, age class and baseline Schirmer I test value as fixed effects and site as random effect; Test type: Superiority — Analysis was based on logistic regression model with multiple imputation (MI) under missing not at random (MNAR) using retrieve dropouts with proportion of patients reaching a value of Schirmer I test >10 mm/5 min at Week 8 as dependent variable, treatment, gender, age class and baseline Schirmer I test value as qualitative independent variables. Site was considered as random effects that vary randomly among patients; p = 0.022, Regression, Logistic; Odds Ratio (OR) = 6.648, 95% CI 2-sided [1.307 to 33.808]

4. Secondary Outcome: Key Secondary Outcome: Change From Baseline in Symptom Assessment in Dry Eye Questionnaire (SANDE) Score for Severity at Week 12
Description: The Symptom Assessment in Dry Eye (SANDE) questionnaire was a short questionnaire to evaluate both dry eye intensity/severity and frequency. This questionnaire used a 100 mm horizontal line (Visual Analogue Scale - VAS) for each of the 2 questions to assess ocular discomfort and/or dryness experienced by the patients. In the SANDE questionnaire, frequency of symptoms ranges from "rarely" to "all of the time" and the severity of symptoms ranged from "very mild" to "very severe". Patients were asked to place a mark on the two given lines based on the extent of their symptoms.
  The locations of the marks was measured in mm from left to right and recorded as frequency and severity scores, respectively.
  The SANDE scale ranged from 0, being the minimal amount of dry eye symptoms (best outcome) to 100, being the maximal amount of dry eye symptoms (worst outcome). In this outcome severity score at week 12 was assessed.
Time Frame: At Week 12 (Visit 5 - Follow-up)
Population: Full Analysis set (FAS): The FAS population consisted of all randomized patients who received at least one dose of the investigational product. The FAS population was used for the primary analysis of the study and to present results on efficacy data.
  While at baseline FAS patients were n=44 for IMP and 40 for Vehicle, at week 4 patients analyzed were n=40 in the IMP group and n=39 in the Vehicle arm.
  Please note that mean is an adjusted mean.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cenegermin - FAS | Vehicle - FAS
Number analyzed (Participants) | 40 | 39
score on a scale | -11.851 [-19.824 to -3.878] | -12.072 [-20.188 to -3.957]
Statistical Analysis 1: Comparison: Cenegermin - FAS vs Vehicle - FAS; Analysis was based on ANCOVA model with multiple imputation (MI) under missing not at random (MNAR) using retrieve dropouts with change from baseline in the severity SANDE score at Week 12 as dependent variable, treatment, gender, age class and baseline severity SANDE score as qualitative independent variables.Site was considered as random effects that vary randomly among patients; Test type: Superiority; p = 0.962, ANCOVA — P-value of adjusted means difference between treatments from the ANCOVA model on change from baseline in SANDE score for severity at Week 12; Adjusted means difference = 0.221, 95% CI 2-sided [-8.934 to 9.377]

5. Secondary Outcome: Key Secondary Outcome: Change From Baseline in Symptoms Assessment in Dry Eye Questionnaire (SANDE) Score for Frequency at Week 12
Description: SANDE was a short questionnaire to evaluate both dry eye intensity and frequency. It uses a 100 mm horizontal line (Visual Analogue Scale, VAS), for each of the 2 questions, to assess ocular discomfort and/or dryness.
  Frequency of symptoms ranged from "rarely" (best outcome) to "all of the time" (worst outcome), while the severity of symptoms ranged from "very mild" (best outcome) to "very severe" (worst outcome). Patients had to place a mark on the two given lines based on the extent of their symptoms.
  The locations of the marks was measured in mm from left to right and recorded as frequency and severity scores, respectively.
  The SANDE lines for intensity and for severity ranged from 0, being the minimal amount of dry eye symptoms (best outcome) to 100, being the maximal amount of dry eye symptoms (worst outcome).
  The total SANDE score was calculated by multiplying the frequency score by the severity score and obtaining the square root (0-100; the lower, the better).
Time Frame: At Week 12 (Visit 5 - Follow-up)
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cenegermin - FAS | Vehicle - FAS
Number analyzed (Participants) | 40 | 39
score on a scale | -14.606 [-23.007 to -6.204] | -14.770 [-23.258 to -6.281]
Statistical Analysis 1: Comparison: Cenegermin - FAS vs Vehicle - FAS; Analysis was based on ANCOVA model with multiple imputation (MI) under missing not at random (MNAR) using retrieve dropouts with change from baseline in the frequency SANDE score at Week 12 as dependent variable, treatment, gender, age class and baseline frequency SANDE score as qualitative independent variables. Site was considered as random effects that vary randomly among patients; Test type: Superiority; p = 0.973, ANCOVA — P-value of adjusted means difference between treatments from the ANCOVA model on change from baseline in SANDE score for frequency at Week 12; Adjusted means difference = 0.164, 95% CI 2-sided [-9.221 to 9.549]

6. Secondary Outcome: Key Secondary Outcome: Change From Baseline in "Quality of Life, Dry Eye Treatment Satisfaction & Bother and Dry Eye Symptom-Bother" Modules Measured by "Impact of Dry Eye on Everyday Life [IDEEL]" Questionnaire at Week 12 and at Week 4.
Description: IDEEL was a 57-item questionnaire that assessed the impact of dry eye symptoms on everyday life. It consisted of 3 modules:
  * Dry eye Quality of Life (27 items) composed by 3 dimensions:
    1. Impact on Daily Activities
    2. Emotional Impact
    3. Impact on Work Scores for each dimension of this module ranged from 0 to 100, where higher scores indicated less impact on daily activities, on work and emotions.
  * Treatment Satisfaction & Bother (8 items) composed by 2 dimensions:
    1. Satisfaction with Treatment Effectiveness
    2. Treatment-Related Bother / Inconvenience Scores for each dimension of this module range from 0 to 100, where higher scores indicate greater satisfaction with treatment effectiveness and less treatment-related bother.
  * Symptom Bother (20 items) composed by 1 dimension:
    1. Dry Eye Symptom-Bother Scores for the dimension of this module ranged from 0 to 100, where higher scores indicated a greater symptom bother.
  No combination of dimensions scores was done.
Time Frame: At Week 12 (Visit 5 - Follow-up) and Week 4 (Visit 3)
Population: Full Analysis set (FAS): it consisted of all randomized patients who received at least one dose of the IMP. The FAS population was used for the primary analysis and to present results on efficacy data. Patients at baseline were n=44 in the cenegermin arm and n=40 in the vehicle arm. At the other timepoints after baseline, a maximum of 43 cenegermin patients and 39 vehicle patients contributed data for this outcome within the FAS population.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cenegermin - FAS | Vehicle - FAS
Number analyzed (Participants) | 43 | 39
score on a scale
  QoL (Daily activities) - Week 4: number analyzed (Participants) | 43 | 38
  QoL (Daily activities) - Week 4 | 13.690 [8.034 to 19.346] | 11.312 [5.393 to 17.231]
  QoL (Daily activities) - Week 12: number analyzed (Participants) | 40 | 38
  QoL (Daily activities) - Week 12 | 13.769 [7.711 to 19.827] | 6.659 [0.549 to 12.769]
  QoL (Feelings) - Week 4 | 8.811 [2.356 to 15.266] | 12.977 [6.263 to 19.692]
  QoL (Feelings) - Week 12: number analyzed (Participants) | 40 | 39
  QoL (Feelings) - Week 12 | 11.413 [5.058 to 17.767] | 10.355 [3.923 to 16.787]
  QoL (Work) - Week 4: number analyzed (Participants) | 27 | 22
  QoL (Work) - Week 4 | 10.689 [2.183 to 19.195] | 14.596 [5.224 to 23.967]
  QoL (Work) - Week 12: number analyzed (Participants) | 27 | 22
  QoL (Work) - Week 12 | 13.225 [5.547 to 20.903] | 13.509 [5.084 to 21.934]
  Treatment Satisfaction (TS) (Treatment - in general) - Week 4: number analyzed (Participants) | 42 | 36
  Treatment Satisfaction (TS) (Treatment - in general) - Week 4 | 8.708 [2.786 to 14.630] | 8.757 [2.493 to 15.022]
  TS (Treatment - in general) - Week 12: number analyzed (Participants) | 39 | 38
  TS (Treatment - in general) - Week 12 | 7.281 [1.570 to 12.992] | 5.305 [-0.513 to 11.124]
  Symptom-Bother - Week 4: number analyzed (Participants) | 43 | 35
  Symptom-Bother - Week 4 | -8.030 [-13.302 to -2.758] | -13.262 [-18.758 to -7.766]
  Symptom-Bother - Week 12: number analyzed (Participants) | 39 | 37
  Symptom-Bother - Week 12 | -10.814 [-16.220 to -5.407] | -10.657 [-16.102 to -5.212]
Statistical Analysis 1: Comparison: Cenegermin - FAS vs Vehicle - FAS; QoL (Daily Activities) - Week 4; Test type: Superiority — Changes from baseline in each IDEEL modules scale score was analyzed using a mixed model for repeated measures (MMRM) adjusting by gender, age class, IDEEL module baseline value, treatment, visit and treatment by visit interaction. Subject was considered as a random effect. The covariance matrix used was "unstructured". Comparisons vs vehicle TID were provided using least square means at each visit and overall; p = 0.52, Mixed Model for Repeated Measures — P-value of LS means difference between treatments from the MMRM on change from baseline in IDEEL Quality of Life Module (Daily Activities) at Week 4; LS means difference = 2.378, 95% CI 2-sided [-4.869 to 9.625]
Statistical Analysis 2: Comparison: Cenegermin - FAS vs Vehicle - FAS; QoL (Daily Activities) - Week 12; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.073, Mixed Model for Repeated Measures — P-value of LS means difference between treatments from the MMRM on change from baseline in IDEEL Quality of Life Module (Daily Activities) at Week 12; LS means difference = 7.11, 95% CI 2-sided [-0.653 to 14.873]
Statistical Analysis 3: Comparison: Cenegermin - FAS vs Vehicle - FAS; QoL (Feelings) - Week 4; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.317, Mixed Model for Repeated Measures — P-value of LS means difference between treatments from the MMRM on change from baseline in IDEEL Quality of Life Module (Feelings) at Week 4; LS means difference = -4.166, 95% CI 2-sided [-12.322 to 3.989]
Statistical Analysis 4: Comparison: Cenegermin - FAS vs Vehicle - FAS; QoL (Feelings) - Week 12; Test type: Superiority — Changes from baseline in each IDEEL modules scale score was analyzed using a mixedmodel for repeated measures (MMRM) adjusting by gender, age class, IDEEL module baseline value, treatment, visit and treatment by visit interaction. Subject was considered as a random effect. The covariance matrix used was "unstructured". Comparisons vs vehicle TID were provided using least square means at each visit and overall; p = 0.792, Mixed Model for Repeated Measures — P-value of LS means difference between treatments from the MMRM on change from baseline in IDEEL Quality of Life Module (Feelings) at Week 12; LS means difference = 1.058, 95% CI 2-sided [-6.786 to 8.901]
Statistical Analysis 5: Comparison: Cenegermin - FAS vs Vehicle - FAS; QoL (Work) - Week 4; Test type: Superiority — Changes from baseline in each IDEEL modules scale score was analyzed using a mixed model for repeated measures (MMRM). Analyses included the fixed, categorical effects of treatment, visit and treatment by visit interaction. Subject was considered as a random effect. The covariance matrix used was "unstructured". Comparisons vs vehicle TID were provided using least square means at each visit and overall. Missing data will be imputed according to the questionnaire manuals; p = 0.488, Mixed Model for Repeated Measures — P-value of LS means difference between treatments from the MMRM on change from baseline in IDEEL Quality of Life Module (Work) at Week 4; LS means difference = -3.907, 95% CI 2-sided [-14.948 to 7.135]
Statistical Analysis 6: Comparison: Cenegermin - FAS vs Vehicle - FAS; QoL (Work) - Week 12; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.954, Mixed Model for Repeated Measures — P-value of LS means difference between treatments from the MMRM on change from baseline in IDEEL Quality of Life Module (Work) at Week 12; LS means difference = -0.284, 95% CI 2-sided [-9.998 to 9.431]
Statistical Analysis 7: Comparison: Cenegermin - FAS vs Vehicle - FAS; TS (Treatment - in general) - Week 4; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.99, Mixed Model for Repeated Measures — P-value of LS means difference between treatments from the MMRM on change from baseline in IDEEL DE Treatment Satisfaction & Bother module (Satisfaction with Treatment Effectiveness) at Week 4; LS means difference = -0.049, 95% CI 2-sided [-7.658 to 7.559]
Statistical Analysis 8: Comparison: Cenegermin - FAS vs Vehicle - FAS; TS (Treatment - in general) - Week 12; Test type: Superiority — Changes from baseline in each IDEEL modules scale score was analyzed using a mixed model for repeated measures (MMRM)adjusting by gender, age class, IDEEL module baseline value, treatment, visit and treatment by visit interaction. Subject was considered as a random effect. The covariance matrix used was "unstructured". Comparisons vs vehicle TID were provided using least square means at each visit and overall; p = 0.582, Mixed Model for Repeated Measures — P-value of LS means difference between treatments from the MMRM on change from baseline in IDEEL DE Treatment Satisfaction & Bother module (Satisfaction with Treatment Effectiveness) at Week 12; LS means difference = 1.976, 95% CI 2-sided [-5.065 to 9.017]
Statistical Analysis 9: Comparison: Cenegermin - FAS vs Vehicle - FAS; Symptom - Bother - Week 4; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.125, Mixed Model for Repeated Measures — P-value of LS means difference between treatments from the MMRM on change from baseline in IDEEL DE Symptom Bother Module at Week 4; LS means difference = 5.232, 95% CI 2-sided [-1.457 to 11.922]
Statistical Analysis 10: Comparison: Cenegermin - FAS vs Vehicle - FAS; Symptom - Bother - Week 12; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.964, Mixed Model for Repeated Measures — P-value of LS means difference between treatments from the MMRM on change from baseline in IDEEL DE Symptom Bother Module at Week 12; LS means difference = -0.156, 95% CI 2-sided [-6.912 to 6.6]

7. Secondary Outcome: Key Secondary Outcome: Change From Baseline in Tear Film Break-Up Time (TFBUT) at Week 4, Week 8 and Week 12
Description: Tear film break-up time (TFBUT) was the time taken to appear first dry spot on cornea after a complete blinking. TFBUT measurement was an easy and fast method used to assess the stability of tear film. It was a standard diagnostic procedure in the dry eye clinics. TFBUT was measured by determining the time to tear break-up. The TFBUT was performed after instillation of 5 μL of 2% preservative-free sodium fluorescein solution into the inferior conjunctival sac of each eye. The patient was instructed to blink several times to thoroughly mix the fluorescein with the tear film.
  A TFBUT greater than 15 seconds was considered normal, while a break time of less than 10 seconds was to be considered pathological. Hence, the shorter the time, the worse the outcome.
Time Frame: At week 4 (Visit 3) , Week 8 (Visit 4), and Week 12 (Visit 5 - Follow-up)
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Cenegermin - FAS | Vehicle - FAS
Number analyzed (Participants) | 43 | 39
seconds
  Week 4 | 1.020 [0.253 to 1.787] | 0.225 [-0.586 to 1.036]
  Week 8: number analyzed (Participants) | 40 | 38
  Week 8 | 0.899 [0.074 to 1.725] | 0.951 [0.088 to 1.813]
  Week 12: number analyzed (Participants) | 40 | 39
  Week 12 | 0.917 [0.123 to 1.711] | 0.782 [-0.040 to 1.603]
Statistical Analysis 1: Comparison: Cenegermin - FAS vs Vehicle - FAS; Analysis was based on MMRM with Multiple Imputation under missing not at random using retrieve dropouts with change from baseline in TFBUT at each timepoint adjusting by gender, age class, TFBUT scale baseline value, treatment, visit, and treatment by visit interaction. Patient was considered as a random effect and the covariance matrix used was unstructured. Herein analysis for Week 4 was reported; Test type: Superiority; p = 0.102, Mixed Model for Repeated Measures — P-value of LS means difference between treatments from the MMRM on change from baseline at Week 4; LS means difference = 0.795, 95% CI 2-sided [-0.157 to 1.748]
Statistical Analysis 2: Comparison: Cenegermin - FAS vs Vehicle - FAS; Analysis was based on MMRM with Multiple Imputation under missing not at random using retrieve dropouts with change from baseline in TFBUT at each timepoint adjusting by gender, age class, TFBUT scale baseline value, treatment, visit, and treatment by visit interaction. Patient was considered as a random effect and the covariance matrix used was unstructured. Herein analysis for Week 8 was reported; Test type: Superiority; p = 0.923, Mixed Model for Repeated Measures — P-value of LS means difference between treatments from the MMRM on change from baseline at Week 8; LS means difference = -0.051, 95% CI 2-sided [-1.094 to 0.991]
Statistical Analysis 3: Comparison: Cenegermin - FAS vs Vehicle - FAS; Analysis was based on MMRM with Multiple Imputation under missing not at random using retrieve dropouts with change from baseline in TFBUT at each timepoint adjusting by gender, age class, TFBUT scale baseline value, treatment, visit, and treatment by visit interaction. Patient was considered as a random effect and the covariance matrix used was unstructured. Herein analysis for Week 12 was reported; Test type: Superiority; p = 0.787, Mixed Model for Repeated Measures — P-value of LS means difference between treatments from the MMRM on change from baseline at Week 12; LS means difference = 0.136, 95% CI 2-sided [-0.849 to 1.12]

8. Secondary Outcome: Change From Baseline in Schirmer I Test (Without Anaesthesia) at Week 4, Week 8, Week 12, and Week 16
Description: The Schirmer test was used in ophthalmic examination to measure tear production for the diagnosis of conditions such as keratoconjunctivitis sicca and dry eye.
  Without previously instilling anesthetic drops, the Schirmer strip was inserted into the lower conjunctival sac at the junction of the lateral and middle thirds, avoiding touching the cornea, and the length of wetting strips in millimeters was recorded after 5 minutes.
  After 5 minutes had elapsed, the Schirmer test strip was removed and the length of the tear absorption on the strip was measured (millimeters/5 minutes).
  Cutoff values:
  <5 mm - pathologic dry eye 5-10 mm - marginal dry eye >10 and <30 mm - normal secretion The longer, the wetted length, the healthier the status of the eye.
Time Frame: At Week 4 (Visit 3), Week 8 (Visit 4), Week 12 (Visit 5), and Week 16 (Visit 6)
Population: Full Analysis set (FAS): it consisted of all randomized patients who received at least one dose of the investigational product. The FAS population was used for the primary analysis of the study and to present results on efficacy data.
  While at baseline FAS patients were n=44 for IMP and 40 for Vehicle, patients analyzed were:
  n=43 at week 4; n=40 at weeks 8 and 12; n=41 at week 16 in the IMP arm and n=39 at weeks 4 and 12; n=40 at weeks 8 and 16 in the vehicle arm.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Cenegermin - FAS | Vehicle - FAS
Number analyzed (Participants) | 43 | 39
millimeters
  Week 4 | 5.4 (5.2) | 1.7 (3.2)
  Week 8: number analyzed (Participants) | 40 | 38
  Week 8 | 4.9 (4.5) | 1.5 (3.0)
  Week 12: number analyzed (Participants) | 40 | 39
  Week 12 | 4.1 (4.7) | 3.1 (6.3)
  Week 16: number analyzed (Participants) | 41 | 38
  Week 16 | 3.4 (4.0) | 2.4 (4.9)
Statistical Analysis 1: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Week 4 (Visit 3) was reported; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — p-value corresponds to a non-parametric Mann-Whitney-Wilcoxon (Wilcoxon rank sum) test of the comparisons between Cenegermin and Vehicle in all patients
Statistical Analysis 2: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Week 8 (Visit 4) was reported; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Week 12 (Visit 5) was reported; Test type: Superiority; p = 0.014, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Week 16 (Visit 6) was reported; Test type: Superiority; p = 0.095, Wilcoxon (Mann-Whitney) — Not statistically significant result. p-value corresponds to a non-parametric Mann-Whitney-Wilcoxon (Wilcoxon rank sum) test of the comparisons between Cenegermin and Vehicle in all patients

9. Secondary Outcome: Change From Baseline in Cornea and Conjunctiva Vital Staining With Fluorescein (National Eye Institute [NEI] Scales) at Week 4, Week 8, Week 12 and Week 16
Description: The NEI/Industry Workshop guidelines were used for grading the scale of corneal and conjunctival damage. The cornea was divided into five sectors (central, superior, inferior, nasal and temporal), each of which was scored on a scale of 0-3, with a maximal total corneal staining score of 15.
  Both nasally and temporally, the conjunctiva was divided into a superior paralimbal area, an inferior paralimbal area, and a peripheral area with a grading scale of 0-3 and with a maximal total score of 9 for the nasal and temporal conjunctiva (overall the total score ranged from 0-18).
  Briefly, grade 0 reflected normal/healthy situation, whereas grade 3 reflected a severe damage in the considered sector.
Time Frame: At Week 4 (Visit 3), Week 8 (Visit 4) , Week 12 (Visit 5) and Week 16 (Visit 6)
Population: Full Analysis set (FAS): it consisted of all randomized patients who received at least one dose of the IMP. The FAS population was used for the primary analysis and to present results on efficacy data. Patients at baseline were n=44 in the cenegermin arm and n=40 in the vehicle arm. At the other timepoints after baseline, a maximum of 42 cenegermin patients and 37 vehicle patients contributed data for this outcome within the FAS population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cenegermin - FAS | Vehicle - FAS
Number analyzed (Participants) | 42 | 37
score on a scale
  corneal and conjunctival damage - Week 4 | -3.6 (4.6) | -2.4 (4.7)
  corneal and conjunctival damage - Week 8: number analyzed (Participants) | 39 | 36
  corneal and conjunctival damage - Week 8 | -3.1 (3.8) | -2.9 (3.9)
  corneal and conjunctival damage - Week 12: number analyzed (Participants) | 39 | 37
  corneal and conjunctival damage - Week 12 | -3.4 (4.6) | -3.0 (3.8)
  corneal and conjunctival damage - Week 16: number analyzed (Participants) | 40 | 36
  corneal and conjunctival damage - Week 16 | -2.0 (6.9) | -2.3 (4.2)
Statistical Analysis 1: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Week 4 (Visit 3) was reported; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Week 8 (Visit 4) was reported; Test type: Superiority; p = 0.328, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Week 12 (Visit 5) was reported; Test type: Superiority; p = 0.287, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Week 16 (Visit 6) was reported; Test type: Superiority; p = 0.777, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]

10. Secondary Outcome: Change From Baseline in Tear Film Break-Up Time (TFBUT) at Week 4, Week 8, Week 12 and Week 16
Description: Tear film break-up time (TFBUT) was the time taken to appear first dry spot on cornea after a complete blinking. TFBUT measurement was an easy and fast method used to assess the stability of tear film. It was a standard diagnostic procedure in the dry eye clinics. TFBUT was measured by determining the time to tear break-up. The TFBUT was performed after instillation of 5 μL of 2% preservative-free sodium fluorescein solution into the inferior conjunctival sac of each eye. The patient was instructed to blink several times to thoroughly mix the fluorescein with the tear film.
  A TFBUT greater than 15 seconds was considered normal, while a break time of less than 10 seconds was to be considered pathological. The shorter the time, the worse the outcome.
Time Frame: At Week 4 (Visit 3), Week 8 (Visit 4), Week 12 (Visit 5), and Week 16 (Visit 6)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cenegermin - FAS | Vehicle - FAS
Number analyzed (Participants) | 43 | 39
seconds
  Week 4 | 1.1 (2.4) | 0.2 (2.2)
  Week 8: number analyzed (Participants) | 40 | 38
  Week 8 | 0.9 (2.5) | 0.9 (2.3)
  Week 12: number analyzed (Participants) | 40 | 39
  Week 12 | 1.0 (2.6) | 0.7 (1.8)
  Week 16: number analyzed (Participants) | 41 | 38
  Week 16 | 1.3 (2.8) | 1.1 (2.5)
Statistical Analysis 1: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Week 4 (Visit 3) was reported; Test type: Superiority; p = 0.126, Wilcoxon (Mann-Whitney) — p-value corresponds to a non-parametric Mann-Whitney-Wilcoxon (Wilcoxon rank sum) test of the comparisons between Cenegermin and and Vehicle in all patients
Statistical Analysis 2: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Week 8 (Visit 4) was reported; Test type: Superiority; p = 0.968, t-test, 2 sided — p-value corresponds to a two sample (independent group) t-test of the comparisons between Cenegermin and Vehicle in all patients
Statistical Analysis 3: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Week 12 (Visit 5) was reported; Test type: Superiority; p = 0.613, t-test, 2 sided — [p-value comment as in outcome 10, analysis 2]
Statistical Analysis 4: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Week 16 (Visit 6) was reported; Test type: Superiority; p = 0.805, t-test, 2 sided — [p-value comment as in outcome 10, analysis 2]

11. Secondary Outcome: Change From Baseline in Symptoms Questionnaire (SANDE) Global Scores, and for Severity and Frequency at Week 8, Week 12, and Week 16
Description: as for outcome 2
Time Frame: At Week 8 (Visit 4), Week 12 (Visit 5), and Week 16 (Visit 6)
Population: Full Analysis set (FAS): it consisted of all randomized patients who received at least one dose of the IMP. The FAS population was used for the primary analysis and to present results on efficacy data. Patients at baseline were n=44 in the cenegermin arm and n=40 in the vehicle arm. At the other timepoints after baseline, a maximum of 41 cenegermin patients and 39 vehicle patients contributed data for this outcome within the FAS population.
  Please note that mean is an adjusted mean.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cenegermin - FAS | Vehicle - FAS
Number analyzed (Participants) | 41 | 39
score on a scale
  Global Score - Week 8: number analyzed (Participants) | 40 | 38
  Global Score - Week 8 | -12.9 (19.0) | -10.3 (19.2)
  Global Score - Week 12: number analyzed (Participants) | 40 | 39
  Global Score - Week 12 | -9.5 (17.0) | -11.3 (22.5)
  Global Score - Week 16: number analyzed (Participants) | 41 | 38
  Global Score - Week 16 | -9.0 (22.3) | -11.1 (19.0)
  Severity - Week 8: number analyzed (Participants) | 40 | 38
  Severity - Week 8 | -10.7 (19.6) | -9.9 (20.9)
  Severity - Week 12: number analyzed (Participants) | 40 | 39
  Severity - Week 12 | -8.6 (19.6) | -10.2 (25.1)
  Severity - Week 16: number analyzed (Participants) | 41 | 38
  Severity - Week 16 | -7.9 (22.9) | -10.2 (20.2)
  Frequency - Week 8: number analyzed (Participants) | 40 | 38
  Frequency - Week 8 | -16.4 (23.2) | -10.9 (21.2)
  Frequency - Week 12: number analyzed (Participants) | 40 | 39
  Frequency - Week 12 | -10.3 (23.6) | -12.3 (23.5)
  Frequency - Week 16: number analyzed (Participants) | 41 | 38
  Frequency - Week 16 | -10.5 (24.2) | -12.2 (18.6)
Statistical Analysis 1: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Global score - Week 8 (Visit 4) was reported; Test type: Superiority; p = 0.543, t-test, 2 sided — p-value corresponds to two sample (independent group) t-test of the comparisons between Cenegermin and Vehicle in all patients
Statistical Analysis 2: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Global score - Week 12 (Visit 5) was reported; Test type: Superiority; p = 0.677, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Global score - Week 16 (Visit 6) was reported; Test type: Superiority; p = 0.914, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Severity - Week 8 (Visit 4) was reported; Test type: Superiority; p = 0.874, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Severity - Week 12 (Visit 5) was reported; Test type: Superiority; p = 0.945, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Severity - Week 16 (Visit 6) was reported; Test type: Superiority; p = 0.727, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 7: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Frequency - Week 8 (Visit 4) was reported; Test type: Superiority; p = 0.342, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 8: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Frequency - Week 12 (Visit 5) was reported; Test type: Superiority; p = 0.821, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 9: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Frequency - Week 16 (Visit 6) was reported; Test type: Superiority; p = 0.926, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]

12. Secondary Outcome: Number of Patients Experienced a Worsening in Symptom Scores (SANDE Global Scores) and/or NEI Score ≥ 50% at Week 4
Description: Symptoms Scores (SANDE) and/or NEI Score were punctually described in the previous outcome descriptions.
  For Sande score, the scale ranges from 0 to 100 for both severity and frequency, where 0 was the best condition and 100 marked the worst condition. Hence the higher the score, the worse the outcome.
  For NEI score, the maximum score (worst outcome) was 15, and the minimum (best outcome) was 0; hence the higher the score, the worse the outcome.
  Please note that mean is an adjusted mean.
Time Frame: At Week 4 (Visit 3)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cenegermin - FAS | Vehicle - FAS
Number analyzed (Participants) | 43 | 39
Participants
  Worsening in symptom scores (SANDE global score) | 14 | 5
  NEI score >= 50%: number analyzed (Participants) | 42 | 37
  NEI score >= 50% | 1 | 1
  Worsening in symptom scores and/or NEI score >= 50: number analyzed (Participants) | 42 | 37
  Worsening in symptom scores and/or NEI score >= 50 | 15 | 5
Statistical Analysis 1: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Worsening in symptom scores (SANDE global score) - Week 4 (Visit 3) was reported; Test type: Superiority; p = 0.0344, Chi-squared — p-value corresponds to Chi-square test of the comparisons between Cenegermin and Vehicle in all patients
Statistical Analysis 2: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for NEI score >= 50% - Week 4 (Visit 3) was reported; Test type: Superiority; p = 1, Fisher Exact — p-value corresponds to a Fisher's exact test of the comparisons between Cenegermin and Vehicle in all patients
Statistical Analysis 3: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Worsening in symptom scores and/or NEI score >= 50 - Week 4 (Visit 3) was reported; Test type: Superiority; p = 0.0235, Chi-squared — p-value corresponds to Chi-square test of the comparisons between Cenegermin and Vehicle in all patients

13. Secondary Outcome: Change From Baseline in "Quality of Life, Dry Eye Treatment Satisfaction & Bother and Dry Eye Symptom-Bother" Modules Measured by "Impact of Dry Eye on Everyday Life [IDEEL]" Questionnaire at Week 4, Week, 8, Week 12, and Week 16
Description: IDEEL was a 57-item questionnaire that assessed the impact of dry eye symptoms on everyday life. It consisted of 3 modules:
  * Dry eye Quality of Life (27 items) composed by 3 dimensions:
    1. Impact on Daily Activities
    2. Emotional Impact
    3. Impact on Work Scores for each dimension of this module ranged from 0 to 100, where higher scores indicated less impact on daily activities, on work and emotions.
  * Treatment Satisfaction & Bother (8 items) composed by 2 dimensions:
    1. Satisfaction with Treatment Effectiveness
    2. Treatment-Related Bother / Inconvenience Scores for each dimension of this module range from 0 to 100, where higher scores indicate greater satisfaction with treatment effectiveness and less treatment-related bother.
  * Symptom Bother (20 items) composed by 1 dimension:
    1. Dry Eye Symptom-Bother. Scores for the dimension of this module ranged from 0 to 100, where higher scores indicated greater symptom bother.
  No combination of dimensions scores was done.
Time Frame: At Week 4 (Visit 3), Week 8 (Visit 4), Week 12 (Visit 5), and Week 16 (Visit 6)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cenegermin - FAS | Vehicle - FAS
Number analyzed (Participants) | 43 | 39
score on a scale
  QoL (Impact on Daily Activities) - Week 4: number analyzed (Participants) | 43 | 38
  QoL (Impact on Daily Activities) - Week 4 | 10.9 (20.7) | 10.3 (16.4)
  QoL (Impact on Daily Activities) - Week 8: number analyzed (Participants) | 40 | 37
  QoL (Impact on Daily Activities) - Week 8 | 9.2 (20.6) | 7.2 (17.0)
  QoL (Impact on Daily Activities) - Week 12: number analyzed (Participants) | 40 | 38
  QoL (Impact on Daily Activities) - Week 12 | 11.9 (20.8) | 5.6 (19.3)
  QoL (Impact on Daily Activities) - Week 16: number analyzed (Participants) | 41 | 37
  QoL (Impact on Daily Activities) - Week 16 | 10.8 (19.6) | 8.1 (16.2)
  QoL (Emotional Impact due to Dry Eye) - Week 4 | 4.3 (21.6) | 10.1 (17.5)
  QoL (Emotional Impact due to Dry Eye) - Week 8: number analyzed (Participants) | 40 | 38
  QoL (Emotional Impact due to Dry Eye) - Week 8 | 6.1 (20.0) | 8.5 (16.0)
  QoL (Emotional Impact due to Dry Eye) - Week 12: number analyzed (Participants) | 40 | 39
  QoL (Emotional Impact due to Dry Eye) - Week 12 | 7.4 (21.8) | 7.4 (16.6)
  QoL (Emotional Impact due to Dry Eye) - Week 16: number analyzed (Participants) | 41 | 38
  QoL (Emotional Impact due to Dry Eye) - Week 16 | 6.7 (25.0) | 7.6 (16.1)
  QoL (Impact on Work due to Dry Eye) - Week 4: number analyzed (Participants) | 27 | 22
  QoL (Impact on Work due to Dry Eye) - Week 4 | 9.8 (24.7) | 13.4 (16.1)
  QoL (Impact on Work due to Dry Eye) - Week 8: number analyzed (Participants) | 28 | 21
  QoL (Impact on Work due to Dry Eye) - Week 8 | 9.5 (21.7) | 8.1 (14.3)
  QoL (Impact on Work due to Dry Eye) - Week 12: number analyzed (Participants) | 27 | 22
  QoL (Impact on Work due to Dry Eye) - Week 12 | 10.4 (19.9) | 11.8 (20.0)
  QoL (Impact on Work due to Dry Eye) - Week 16: number analyzed (Participants) | 28 | 22
  QoL (Impact on Work due to Dry Eye) - Week 16 | 13.6 (21.3) | 8.9 (15.1)
  TS (Satisfaction with Effectiveness) - Week 4: number analyzed (Participants) | 42 | 36
  TS (Satisfaction with Effectiveness) - Week 4 | 11.3 (30.4) | 10.1 (25.1)
  TS (Satisfaction with Effectiveness) - Week 8: number analyzed (Participants) | 39 | 37
  TS (Satisfaction with Effectiveness) - Week 8 | 12.0 (25.5) | 5.2 (25.2)
  TS (Satisfaction with Effectiveness) - Week 12: number analyzed (Participants) | 39 | 38
  TS (Satisfaction with Effectiveness) - Week 12 | 13.1 (26.8) | 7.4 (25.7)
  TS (Satisfaction with Effectiveness) - Week 16: number analyzed (Participants) | 40 | 37
  TS (Satisfaction with Effectiveness) - Week 16 | 13.1 (29.0) | 7.9 (26.1)
  TS (Treatment Bother/Inconvenience) - Week 4: number analyzed (Participants) | 43 | 35
  TS (Treatment Bother/Inconvenience) - Week 4 | 5.5 (21.7) | 6.2 (12.7)
  TS (Treatment Bother/Inconvenience) - Week 8: number analyzed (Participants) | 39 | 36
  TS (Treatment Bother/Inconvenience) - Week 8 | 3.3 (18.9) | 5.0 (14.8)
  TS (Treatment Bother/Inconvenience) - Week 12: number analyzed (Participants) | 39 | 37
  TS (Treatment Bother/Inconvenience) - Week 12 | 4.5 (19.8) | 4.2 (12.4)
  TS (Treatment Bother/Inconvenience) - Week 16: number analyzed (Participants) | 39 | 36
  TS (Treatment Bother/Inconvenience) - Week 16 | 5.4 (18.5) | 3.3 (11.3)
  Symptom-Bother - Week 4 | -5.8 (18.7) | -11.9 (12.5)
  Symptom-Bother - Week 8: number analyzed (Participants) | 40 | 38
  Symptom-Bother - Week 8 | -7.2 (16.4) | -7.9 (12.9)
  Symptom-Bother - Week 12: number analyzed (Participants) | 40 | 39
  Symptom-Bother - Week 12 | -8.6 (15.5) | -9.5 (17.7)
  Symptom-Bother - Week 16: number analyzed (Participants) | 41 | 38
  Symptom-Bother - Week 16 | -8.0 (17.0) | -9.2 (13.9)
Statistical Analysis 1: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for QoL (Impact on Daily Activities) - Week 4 (Visit 3) was reported; Test type: Superiority; p = 0.888, t-test, 2 sided — [p-value comment as in outcome 10, analysis 2]
Statistical Analysis 2: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for QoL (Impact on Daily Activities) - Week 8 (Visit 4) was reported; Test type: Superiority; p = 0.651, t-test, 2 sided — [p-value comment as in outcome 10, analysis 2]
Statistical Analysis 3: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for QoL (Impact on Daily Activities) - Week 12 (Visit 5) was reported; Test type: Superiority; p = 0.267, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for QoL (Impact on Daily Activities) - Week 16 (Visit 6) was reported; Test type: Superiority; p = 0.459, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for QoL (Emotional Impact due to Dry Eye) - Week 4 was reported; Test type: Superiority; p = 0.192, t-test, 2 sided — [p-value comment as in outcome 10, analysis 2]
Statistical Analysis 6: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for QoL (Emotional Impact due to Dry Eye) - Week 8 was reported; Test type: Superiority; p = 0.568, t-test, 2 sided — [p-value comment as in outcome 10, analysis 2]
Statistical Analysis 7: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for QoL (Emotional Impact due to Dry Eye) - Week 12 was reported; Test type: Superiority; p = 0.871, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 8: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for QoL (Emotional Impact due to Dry Eye) - Week 16 was reported; Test type: Superiority; p = 0.85, t-test, 2 sided — [p-value comment as in outcome 10, analysis 2]
Statistical Analysis 9: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for QoL (Impact on Work due to Dry Eye) - Week 4 was reported; Test type: Superiority; p = 0.364, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 10: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for QoL (Impact on Work due to Dry Eye) - Week 8 was reported; Test type: Superiority; p = 0.646, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 11: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for QoL (Impact on Work due to Dry Eye) - Week 12 was reported; Test type: Superiority; p = 0.739, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 12: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for QoL (Impact on Work due to Dry Eye) - Week 16 was reported; Test type: Superiority; p = 0.664, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 13: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for TS (Satisfaction with Effectiveness) - Week 4 was reported; Test type: Superiority; p = 0.846, t-test, 2 sided — [p-value comment as in outcome 10, analysis 2]
Statistical Analysis 14: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for TS (Satisfaction with Effectiveness) - Week 8 was reported; Test type: Superiority; p = 0.248, t-test, 2 sided — [p-value comment as in outcome 10, analysis 2]
Statistical Analysis 15: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for TS (Satisfaction with Effectiveness) - Week 12 was reported; Test type: Superiority; p = 0.341, t-test, 2 sided — [p-value comment as in outcome 10, analysis 2]
Statistical Analysis 16: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for TS (Satisfaction with Effectiveness) - Week 16 was reported; Test type: Superiority; p = 0.413, t-test, 2 sided — [p-value comment as in outcome 10, analysis 2]
Statistical Analysis 17: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for TS (Treatment Bother/Inconvenience) - Week 4 was reported; Test type: Superiority; p = 0.927, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 18: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for TS (Treatment Bother/Inconvenience) - Week 8 was reported; Test type: Superiority; p = 0.914, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 19: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for TS (Treatment Bother/Inconvenience) - Week 12 was reported; Test type: Superiority; p = 0.564, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 20: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for TS (Treatment Bother/Inconvenience) - Week 16 was reported; Test type: Superiority; p = 0.489, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 21: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Symptom-Bother - Week 4; Test type: Superiority; p = 0.082, t-test, 2 sided — [p-value comment as in outcome 10, analysis 2]
Statistical Analysis 22: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Symptom-Bother - Week 8 was reported; Test type: Superiority; p = 0.848, t-test, 2 sided — [p-value comment as in outcome 10, analysis 2]
Statistical Analysis 23: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Symptom-Bother - Week 12 was reported; Test type: Superiority; p = 0.805, t-test, 2 sided — [p-value comment as in outcome 10, analysis 2]
Statistical Analysis 24: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Symptom-Bother - Week 16 was reported; Test type: Superiority; p = 0.833, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]

14. Other Pre Specified Outcome: Number of Patients With at Least One Treatment-emergent Adverse Event (TEAE) From Screening Day to Week 24
Description: Treatment emergent adverse events (TEAEs) were undesirable events not present prior to medical treatment, or an already present event that worsens either in intensity or frequency following the treatment.
Time Frame: From Screening day (Day -8) up to Week 24 (Visit 7 - Follow-up)
Population: The SAF set consisted of all randomized patients who received at least one dose of the investigational product. SAF set was analyzed according to the actual treatment received. The SAF population was used to present results on safety data.
Measure: Count of Participants; unit: Participants
Groups:
- Cenegermin - SAF: One drop of cenegermin 20 mcg/mL (rhNGF 20 mcg/mL), in the pharmaceutical form of ophthalmic sterile solution, was instilled in both eyes three times daily (TID), every six hours.
  Cenegermin: Oxervate®, an ophthalmic solution containing cenegermin 20 mcg/mL, which is a recombinant human Nerve Growth Factor (rhNGF); one drop of the test product will be instilled in both eyes three times daily (TID).
- Vehicle - SAF: In this arm one drop of vehicle was instilled in both eyes TID for 28 consecutive days.
  Vehicle: Vehicle was instilled with the same scheme of the test product
Arm/Group | Cenegermin - SAF | Vehicle - SAF
Number analyzed (Participants) | 44 | 40
Participants
  Any TEAE | 27 | 18
  Any TEAE - Ophtalmic | 26 | 12
  Any TEAE . Non-ophtalmic | 9 | 9
  Any severe TEAE | 0 | 1
  Any severe TEAE - Ophtalmic | 0 | 1
  Any severe TEAE - Non-ophtalmic | 0 | 0
  Any serious TEAE | 0 | 0
  Any serious TEAE - Ophtalmic | 0 | 0
  Any serious TEAE - Non-ophtalmic | 0 | 0
  Any non-serious TEAE | 27 | 18
  Any ADR | 26 | 12
  Any ADR - Ophtalmic | 26 | 10
  Any ADR - Non-ophtalmic | 3 | 4
  Any Serious ADR | 0 | 0
  Any Serious ADR leading to IMP discontinuation | 0 | 1
  Any TEAE leading to study discontinuation | 0 | 1
  Any TEAE leading to death | 0 | 0

15. Other Pre Specified Outcome: Use of Preservative Free Artificial Tears Use (Number of Drops/Day).
Description: Use of Preservative Free Artificial Tears by Study Period is calculated as: total number of drops of the preservative free artificial tears during the X period/ total number of days of the X period * 100.
Time Frame: Treatment period (Day 1 to Week 4), Follow-up period (Week 4 to Week 24), Overall period (Day 1 to Week 24)
Population: Full Analysis set (FAS): it consisted of all randomized patients who received at least one dose of the IMP. The FAS population was used for the primary analysis and to present results on efficacy data. Patients at baseline were n=44 in the cenegermin arm and n=40 in the vehicle arm. At the other timepoints after baseline, a maximum of 41 cenegermin patients and 38 vehicle patients contributed data for this outcome within the FAS population.
Measure: Median (Standard Deviation); unit: number of drops
Arm/Group | Cenegermin - FAS | Vehicle - FAS
Number analyzed (Participants) | 41 | 38
number of drops
  Treatment period: number analyzed (Participants) | 40 | 35
  Treatment period | 261.2 (220.2) | 215.7 (184.7)
  Follow-up period: number analyzed (Participants) | 38 | 37
  Follow-up period | 330.0 (178.1) | 317.6 (168.3)
  Overall period | 294.7 (202.5) | 268.1 (182.6)

16. Other Pre Specified Outcome: Change From Baseline in Schirmer I Test (Without Anaesthesia) at Week 2
Description: as for outcome 8
Time Frame: At week 2 (Visit 2)
Population: Full Analysis set (FAS): The FAS population consisted of all randomized patients who received at least one dose of the investigational product.
  While at baseline FAS patients were n=44 for IMP and 40 for Vehicle, at week 2 patients analyzed were n=43 in the IMP group and n=39 in the Vehicle arm.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Cenegermin - FAS | Vehicle - FAS
Number analyzed (Participants) | 43 | 39
millimeters | 4.4 (5.0) | 1.0 (2.4)
Statistical Analysis 1: Comparison: Cenegermin - FAS vs Vehicle - FAS; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]

17. Other Pre Specified Outcome: Change From Baseline in Cornea and Conjunctiva Vital Staining With Fluorescein (National Eye Institute [NEI] Scales) at Week 2
Description: as for outcome 9
Time Frame: At Week 2 (Visit 2)
Population: Full Analysis set (FAS): The FAS population consisted of all randomized patients who received at least one dose of the investigational product. FAS population was analysed according to intention-to-treat (ITT) principle, i.e., by treatment allocation regardless happening of intercurrent events (treatment policy strategy).
  Herein the Number Participants Analyzed in Cenergermin group was 42, in the Vehicle group was 37.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cenegermin - FAS | Vehicle - FAS
Number analyzed (Participants) | 42 | 37
score on a scale | -2.6 (4.8) | -2.0 (5.2)
Statistical Analysis 1: Comparison: Cenegermin - FAS vs Vehicle - FAS; Test type: Superiority; p = 0.046, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]

18. Other Pre Specified Outcome: Change From Baseline in Tear Film Break-Up Time (TFBUT) at Week 2
Description: Tear film break-up time (TFBUT) was the time taken to appear first dry spot on cornea after a complete blinking. TFBUT measurement was an easy and fast method used to assess the stability of tear film. It was a standard diagnostic procedure in the dry eye clinics. TFBUT was measured by determining the time to tear break-up. The TFBUT was performed after instillation of 5 μL of 2% preservative-free sodium fluorescein solution into the inferior conjunctival sac of each eye. The patient was instructed to blink several times to thoroughly mix the fluorescein with the tear film.
  A TFBUT greater than 15 seconds was considered normal, while a break time of less than 10 seconds was to be considered pathological.
Time Frame: At Week 2 (Visit 2)
Population: Full Analysis set (FAS): The FAS population consisted of all randomized patients who received at least one dose of the investigational product. FAS population was analysed according to intention-to-treat (ITT) principle, i.e., by treatment allocation regardless happening of intercurrent events (treatment policy strategy).
  Herein the Number Participants Analyzed in Cenergermin group was 43, in the Vehicle group was 39.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cenegermin - FAS | Vehicle - FAS
Number analyzed (Participants) | 43 | 39
seconds | 0.7 (2.1) | 0.2 (2.0)
Statistical Analysis 1: Comparison: Cenegermin - FAS vs Vehicle - FAS; Test type: Superiority; p = 0.34, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]

19. Other Pre Specified Outcome: Change From Baseline in Symptoms Questionnaire (SANDE) Global Scores, and for Severity and Frequency at Week 2, and Week 4
Description: as for outcome 2
Time Frame: At Week 2 (Visit 2) and Week 4 (Visit 3)
Population: Full Analysis set (FAS): it consisted of all randomized patients who received at least one dose of the IMP. The FAS population was used for the primary analysis and to present results on efficacy data. Patients at baseline were n=44 in the cenegermin arm and n=40 in the vehicle arm. At the other timepoints after baseline, only 43 cenegermin patients and 39 vehicle patients contributed data for this outcome within the FAS population.
  Please note that mean is an adjusted mean.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cenegermin - FAS | Vehicle - FAS
Number analyzed (Participants) | 43 | 39
score on a scale
  Global Score - Change from baseline to Week 2 | -2.1 (18.0) | -12.3 (13.7)
  Global Score - Change from baseline to Week 4 | -11.5 (17.4) | -15.0 (18.0)
  Severity - Change from baseline to Week 2 | -0.5 (20.1) | -12.3 (14.9)
  Severity - Change from baseline to Week 4 | -9.2 (19.7) | -13.6 (17.2)
  Frequency - Change from baseline to Week 2 | -3.8 (18.9) | -12.0 (14.7)
  Frequency - Change from baseline to Week 4 | -14.5 (18.8) | -16.9 (22.2)
Statistical Analysis 1: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Global Score - Week 2 was reported; Test type: Superiority; p = 0.017, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Global Score - Week 4 was reported; Test type: Superiority; p = 0.339, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Severity - Week 2 was reported; Test type: Superiority; p = 0.004, t-test, 2 sided — [p-value comment as in outcome 10, analysis 2]
Statistical Analysis 4: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Severity - Week 4 was reported; Test type: Superiority; p = 0.292, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Frequency - Week 2 was reported; Test type: Superiority; p = 0.09, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Frequency - Week 4 was reported; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]

20. Other Pre Specified Outcome: Number of Patients Experienced a Worsening in Symptom Scores (SANDE Global Score) and/or NEI Score ≥ 50% Assessed at Week 2
Description: Symptoms Scores (SANDE) and/or NEI Score were punctually described in the previous outcome descriptions.
  For Sande score, the scale ranges from 0 to 100 for both severity and frequency, where 0 was the best condition and 100 marked the worst condition. Hence the higher the score, the worse the outcome.
  For NEI score, the maximum score (worst outcome) was 15, and the minimum (best outcome) was 0; hence the higher the score, the worse the outcome.
Time Frame: At Week 2 (Visit 2)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cenegermin - FAS | Vehicle - FAS
Number analyzed (Participants) | 43 | 39
Participants
  Worsening in symptom scores (SANDE global score) | 17 | 5
  NEI score >= 50%: number analyzed (Participants) | 42 | 37
  NEI score >= 50% | 1 | 0
  Worsening in symptom scores and/or NEI score >= 50: number analyzed (Participants) | 42 | 38
  Worsening in symptom scores and/or NEI score >= 50 | 18 | 5
Statistical Analysis 1: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Worsening in symptom scores (SANDE global score) was reported; Test type: Superiority; p = 0.0064, Chi-squared — p-value corresponds to Chi-square test of the comparisons between Cenegermin and Vehicle in all patients
Statistical Analysis 2: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for NEI score >= 50% was reported; Test type: Superiority; p = 1, Fisher Exact — p-value corresponds to a Fisher's exact test of the comparisons between Cenegermin and Vehicle in all patients
Statistical Analysis 3: Comparison: Cenegermin - FAS vs Vehicle - FAS; Herein analysis for Worsening in symptom scores and/or NEI score >= 50 was reported; Test type: Superiority; p = 0.0034, Chi-squared — p-value corresponds to Chi-square test of the comparisons between Cenegermin and Vehicle in all patients

21. Other Pre Specified Outcome: Change From Baseline in Schirmer Test II (With Topical Anaesthesia) at Week 4
Description: Schirmer Test II (with anaesthetic) measured baseline plus reflex secretion. The Schirmer strip was inserted into the lower conjunctival sac at the junction of the lateral and middle thirds, avoiding touching the cornea, and the length of wetting strips in millimeters was recorded after 5 minutes.
  After 5 minutes had elapsed, the Schirmer test strip was removed and the length of the tear absorption on the strip was measured (millimeters/5 minutes).
  Cutoff values:
  <5 mm - pathologic dry eye 5-10 mm - marginal dry eye >10 and <30 mm - normal secretion The longer, the wetted length, the healthier the status of the eye.
Time Frame: At Week 4 (Visit 3)
Population: Full Analysis set (FAS): The FAS population consisted of all randomized patients who received at least one dose of the investigational product.
  While at baseline FAS patients were n=44 for IMP and 40 for Vehicle, at week 4 patients analyzed were n=42 in the IMP group and n=38 in the Vehicle arm.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Cenegermin - FAS | Vehicle - FAS
Number analyzed (Participants) | 42 | 38
millimeters | 4.3 (4.2) | 1.4 (3.7)
Statistical Analysis 1: Comparison: Cenegermin - FAS vs Vehicle - FAS; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — p-value corresponds to a non-parametric Mann-Whitney-Wilcoxon (Wilcoxon rank sum) test of the comparisons between Cenegermin and Vehicle in all participants

22. Other Pre Specified Outcome: Change From Baseline in Best Corrected Distance Visual Acuity (BCDVA)
Description: Best corrected visual acuity (BCDVA) was determined by careful refraction according to the standard protocol for refraction. Chart 1 was used for testing the VA of the right eye; Chart 2 for the left eye; and Chart R for refraction only.
  Retroilluminated standard Early Treatment of Diabetic Retinopathy Study (ETDRS) charts were used. They had 5 Sloan letters on each line of equal difficulty, and there was a geometric progression in letter size from line to line. VAS awarded one point for every letter correctly guessed. A distance of 4 meters was required between the subject's eyes and the VA chart. When a subject cannot read at least 20 letters on the chart at 4 meters, the subject was tested at 1 meter. If 20 or more letters were read at 4 meters, the VAS for that eye was recorded as the number of letters correct at 4 meters plus 30. Otherwise, the VAS was the number of letters read correctly at 1 meter plus the number read at 4 meters. The higher the score the better the outcome.
Time Frame: At Week 2 (Visit 2), Week 4 (Visit 3), Week 8 (Visit 4), Week 12 (Visit 5), and Week 16 (Visit 6)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cenegermin - FAS | Vehicle - FAS
Number analyzed (Participants) | 43 | 39
Participants
  CFB to Week 2 - No change | 32 | 29
  CFB to Week 2 - 20/63 to 20/40 | 0 | 1
  CFB to Week 2 - 20/50 to 20/40 | 0 | 1
  CFB to Week 2 - 20/40 to 20/25 | 1 | 1
  CFB to Week 2 - 20/32 to 20/20 | 1 | 0
  CFB to Week 2 - 20/32 to 20/25 | 1 | 1
  CFB to Week 2 - 20/25 to 20/20 | 3 | 2
  CFB to Week 2 - 20/20 to 20/16 | 2 | 0
  CFB to Week 2 - 20/20 to 20/25 | 1 | 2
  CFB to Week 2 - 20/16 to 20/12.5 | 0 | 1
  CFB to Week 2 - 20/16 to 20/20 | 1 | 0
  CFB to Week 2 - 20/16 to 20/25 | 1 | 0
  CFB to Week 2 - 20/16 to 20/32 | 0 | 1
  CFB to Week 4 - No change | 31 | 33
  CFB to Week 4 - 20/63 to 20/40 | 0 | 1
  CFB to Week 4 - 20/40 to 20/25 | 1 | 1
  CFB to Week 4 - 20/40 to 20/32 | 1 | 0
  CFB to Week 4 - 20/32 to 20/20 | 0 | 1
  CFB to Week 4 - 20/32 to 20/25 | 1 | 0
  CFB to Week 4 - 20/25 to 20/20 | 3 | 2
  CFB to Week 4 - 20/20 to 20/25 | 3 | 0
  CFB to Week 4 - 20/20 to 20/32 | 1 | 0
  CFB to Week 4 - 20/16 to 20/20 | 2 | 0
  CFB to Week 4 - 20/16 to 20/32 | 0 | 1
  CFB to Week 8 - No change: number analyzed (Participants) | 40 | 38
  CFB to Week 8 - No change | 26 | 29
  CFB to Week 8 - 20/63 to 20/40: number analyzed (Participants) | 40 | 38
  CFB to Week 8 - 20/63 to 20/40 | 0 | 1
  CFB to Week 8 - 20/50 to 20/40: number analyzed (Participants) | 40 | 38
  CFB to Week 8 - 20/50 to 20/40 | 0 | 1
  CFB to Week 8 - 20/40 to 20/20: number analyzed (Participants) | 40 | 38
  CFB to Week 8 - 20/40 to 20/20 | 0 | 1
  CFB to Week 8 -20/40 to 20/25: number analyzed (Participants) | 40 | 38
  CFB to Week 8 -20/40 to 20/25 | 1 | 0
  CFB to Week 8 -20/40 to 20/32: number analyzed (Participants) | 40 | 38
  CFB to Week 8 -20/40 to 20/32 | 1 | 0
  CFB to Week 8 - 20/40 to 20/50: number analyzed (Participants) | 40 | 38
  CFB to Week 8 - 20/40 to 20/50 | 1 | 0
  CFB to Week 8 -20/32 to 20/20: number analyzed (Participants) | 40 | 38
  CFB to Week 8 -20/32 to 20/20 | 1 | 0
  CFB to Week 8 -20/32 to 20/25: number analyzed (Participants) | 40 | 38
  CFB to Week 8 -20/32 to 20/25 | 1 | 1
  CFB to Week 8 - 20/25 to 20/20: number analyzed (Participants) | 40 | 38
  CFB to Week 8 - 20/25 to 20/20 | 2 | 1
  CFB to Week 8 - 20/25 to 20/32: number analyzed (Participants) | 40 | 38
  CFB to Week 8 - 20/25 to 20/32 | 1 | 0
  CFB to Week 8 - 20/20 to 20/16: number analyzed (Participants) | 40 | 38
  CFB to Week 8 - 20/20 to 20/16 | 2 | 1
  CFB to Week 8 - 20/20 to 20/25: number analyzed (Participants) | 40 | 38
  CFB to Week 8 - 20/20 to 20/25 | 2 | 2
  CFB to Week 8 - 20/16 to 20/20: number analyzed (Participants) | 40 | 38
  CFB to Week 8 - 20/16 to 20/20 | 2 | 0
  CFB to Week 8 -20/16 to 20/32: number analyzed (Participants) | 40 | 38
  CFB to Week 8 -20/16 to 20/32 | 0 | 1
  CFB to Week 12 - no change: number analyzed (Participants) | 40 | 39
  CFB to Week 12 - no change | 29 | 30
  CFB to Week 12 - 20/63 to 20/80: number analyzed (Participants) | 40 | 39
  CFB to Week 12 - 20/63 to 20/80 | 0 | 1
  CFB to Week 12 -20/50 to 20/63: number analyzed (Participants) | 40 | 39
  CFB to Week 12 -20/50 to 20/63 | 0 | 1
  CFB to Week 12 -20/40 to 20/20: number analyzed (Participants) | 40 | 39
  CFB to Week 12 -20/40 to 20/20 | 0 | 1
  CFB to Week 12 - 20/40 to 20/32: number analyzed (Participants) | 40 | 39
  CFB to Week 12 - 20/40 to 20/32 | 1 | 0
  CFB to Week 12 - 20/32 to 20/20: number analyzed (Participants) | 40 | 39
  CFB to Week 12 - 20/32 to 20/20 | 1 | 0
  CFB to Week 12 - 20/32 to 20/25: number analyzed (Participants) | 40 | 39
  CFB to Week 12 - 20/32 to 20/25 | 1 | 1
  CFB to Week 12 - 20/25 to 20/20: number analyzed (Participants) | 40 | 39
  CFB to Week 12 - 20/25 to 20/20 | 3 | 1
  CFB to Week 12 - 20/25 to 20/32: number analyzed (Participants) | 40 | 39
  CFB to Week 12 - 20/25 to 20/32 | 1 | 0
  CFB to Week 12 - 20/20 to 20/16: number analyzed (Participants) | 40 | 39
  CFB to Week 12 - 20/20 to 20/16 | 0 | 1
  CFB to Week 12 -20/20 to 20/25: number analyzed (Participants) | 40 | 39
  CFB to Week 12 -20/20 to 20/25 | 1 | 2
  CFB to Week 12 - 20/20 to 20/32: number analyzed (Participants) | 40 | 39
  CFB to Week 12 - 20/20 to 20/32 | 1 | 0
  CFB to Week 12 -20/16 to 20/20: number analyzed (Participants) | 40 | 39
  CFB to Week 12 -20/16 to 20/20 | 1 | 0
  CFB to Week 12 -20/16 to 20/50: number analyzed (Participants) | 40 | 39
  CFB to Week 12 -20/16 to 20/50 | 0 | 1
  CFB to Week 12 - 20/12.5 to 20/16: number analyzed (Participants) | 40 | 39
  CFB to Week 12 - 20/12.5 to 20/16 | 1 | 0
  CFB to Week 16 - no change: number analyzed (Participants) | 41 | 38
  CFB to Week 16 - no change | 25 | 27
  CFB to Week 16 -20/63 to 20/50: number analyzed (Participants) | 41 | 38
  CFB to Week 16 -20/63 to 20/50 | 0 | 1
  CFB to Week 16 -20/50 to 20/40: number analyzed (Participants) | 41 | 38
  CFB to Week 16 -20/50 to 20/40 | 0 | 1
  CFB to Week 16 - 20/40 to 20/20: number analyzed (Participants) | 41 | 38
  CFB to Week 16 - 20/40 to 20/20 | 0 | 1
  CFB to Week 16 -20/40 to 20/25: number analyzed (Participants) | 41 | 38
  CFB to Week 16 -20/40 to 20/25 | 1 | 0
  CFB to Week 16 -20/40 to 20/32: number analyzed (Participants) | 41 | 38
  CFB to Week 16 -20/40 to 20/32 | 1 | 0
  CFB to Week 16 - 20/40 to 20/50: number analyzed (Participants) | 41 | 38
  CFB to Week 16 - 20/40 to 20/50 | 1 | 0
  CFB to Week 16 -20/32 to 20/25: number analyzed (Participants) | 41 | 38
  CFB to Week 16 -20/32 to 20/25 | 2 | 2
  CFB to Week 16 -20/25 to 20/16: number analyzed (Participants) | 41 | 38
  CFB to Week 16 -20/25 to 20/16 | 0 | 1
  CFB to Week 16 -20/25 to 20/20: number analyzed (Participants) | 41 | 38
  CFB to Week 16 -20/25 to 20/20 | 4 | 0
  CFB to Week 16 -20/25 to 20/32: number analyzed (Participants) | 41 | 38
  CFB to Week 16 -20/25 to 20/32 | 0 | 2
  CFB to Week 16 -20/20 to 20/16: number analyzed (Participants) | 41 | 38
  CFB to Week 16 -20/20 to 20/16 | 3 | 0
  CFB to Week 16 -20/20 to 20/25: number analyzed (Participants) | 41 | 38
  CFB to Week 16 -20/20 to 20/25 | 2 | 2
  CFB to Week 16 -20/16 to 20/20: number analyzed (Participants) | 41 | 38
  CFB to Week 16 -20/16 to 20/20 | 2 | 1

ADVERSE EVENTS:
Time Frame: AEs were collected from the screening visit (Day -8) until last Follow-Up visit (Week 24).
Description: An AE was defined as any untoward medical occurrence in a patient or clinical investigation patient administered a medicinal product and which did not necessarily have a causal relationship with this treatment. Please note that analyses in NGF0221 were done at the patient level, not by eye, so adverse events reported may refer to the study eye, the non-study eye, or both, indifferently.
Arm/Group | Cenegermin - SAF | Vehicle - SAF
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/40
Other Adverse Events (participants affected / at risk) | 27/44 | 18/40
OTHER ADVERSE EVENTS (reported when occurring in more than 4.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cenegermin - SAF (N=44) | Vehicle - SAF (N=40)
Conjunctival hyperaemia (Eye disorders) | 2 (2) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 3 (3)
Eye discharge (Eye disorders) | 2 (2) | 2 (3)
Eye irritation (Eye disorders) | 2 (2) | 1 (1)
Eye pain (Eye disorders) | 21 (23) | 4 (4)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 2 (2)
Photophobia (Eye disorders) | 2 (2) | 0 (0)
Swelling of eyelid (Eye disorders) | 2 (2) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 2 (2)
Eyelid pain (Eye disorders) | 7 (9) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT05136170/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/70/NCT05136170/SAP_001.pdf